CLINICAL TRIAL: NCT03725566
Title: Phase I Clinical Trial of Recombinant Humanized Anti-vegf Monoclonal Antibody Single Vitreous Injection for Safety, Tolerance, PK and Pharmacodynamics in nAMD Patients
Brief Title: JY028 Single Vitreous Injection in a Phase 1 Clinical Trial in nAMD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2017L02087
Record Dates: First submitted 2018-09-20; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-09

CONDITIONS: Macular Degeneration
Keywords: New vascular macular degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental (Experimental): Recombinant humanized anti-VEGF monoclonal antibody injection 0.625mg/1.25mg/2.0mg/2.5mg by intravitreous injection,day 1 in the first month;
  Interventions: Drug: Experimental

INTERVENTIONS:
Drug: Experimental — Recombinant humanized anti-VEGF monoclonal antibody injection 0.625mg/1.25mg/2.0mg/2.5mg by intravitreous injection,day 1 in the first month;
  Other Names: intravitreous injection

SUMMARY:
Phase I clinical trial on safety, tolerance, pharmacokinetics (PK) and pharmacodynamics of recombinant human anti-VEGF monoclonal antibody injection in patients with neovascular (wet) age-related macular degeneration

DETAILED DESCRIPTION:
Test drug:Recombinant humanized anti VEGF monoclonal antibody injection; Research Phase:Phase I; Subjects:Subjects with neovascular (wet) age-related macular degeneration; Number of Subjects:24; Trial design:Single center, non randomized, open, single arm, single dose, dose escalation; Research objective:to rearch the safety and tolerance of JY028 injection;to rearch PK of JY028 injection;to observe the efficacy of JY028 in the treatment of nAMD;to rearch the relationship between plasma VEGF concentration and JY028 concentration. to rearch immunogenicity of JY028;

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteered to participate and signed the informed consent 2. No more than 50 years of age and less than 75 years of age, male or female 3. Diagnosed as nAMD 4. The optimal corrected visual acuity of the target eye ETDRS should be no more than 50 letters, and the optimal corrected visual acuity of the opposite eye should be no more than 34 letters 5. The target eye pressure is no more than 25mmHg, which can be controlled by drugs 6. A normal coagulation function: the platelet count is 100 x 10 ^ 9-300x 10^10 / L, thrombin time, prothrombin time within the normal range.

-

Exclusion Criteria:

1. Choroid polypoid angiopathy (PCV)
2. There are other obvious eye diseases/conditions (such as diabetic retinopathy, cataract, abnormal eyelid, uncontrolled glaucoma, eye active inflammation, etc.)
3. CNV caused by other causes other than nAMD, such as diabetic retinopathy, vascular stripe disease, ocular histoplasmosis, case myopia, trauma, etc
4. The target eye has received any intraocular surgery or laser therapy within 3 months prior to enrollment
5. Any eye treated with antiangiogenic drugs within 3 months prior to baseline visit
6. Patients with active eye infections, such as conjunctivitis, keratitis, sclerotic, blepharitis, endophthalmitis or uveitis
7. Persons with a history of myocardial infarction and/or cerebral infarction or other active or acute cardiovascular diseases
8. HIV antibody/hiv-p24 antigen, any of the positive subjects in the treponema pallidum antibody
9. Active HBsAg carriers (conditions must be met: HBsAg positive, HBV DNA positive, ALT higher than normal upper limit)
10. Patients with HCV (the following conditions must be met: lgM positive anti-hcv antibody, ALT higher than the upper limit of normal value)
11. Fluorescein sodium allergy
12. Allergy to anti-vegf monoclonal antibodies or humanized monoclonal antibodies
13. Patients who participated in other clinical trials within 3 months
14. Patients who took NSAIDs and aspirin or other anticoagulant or platelet drugs within 1 month before enrollment
15. An unhealed wound, ulcer, fracture, or other related medical condition
16. Patients with uncontrollable hypertension, with systolic blood pressure of > 140mmHg and diastolic blood pressure of > 90mmHg
17. Patients with uncontrollable clinical diseases or problems (such as serious mental, neurological, cardiovascular, respiratory and other systemic diseases and malignant tumors)
18. Pregnant and lactating women and those who cannot take contraceptive measures
19. According to the researcher, it is not suitable for the candidate -

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
JY028 related incidence of ocular and systemic adverse events and serious adverse events | 13 weeks
  JY028 related incidence of ocular and systemic adverse events and serious adverse events

SECONDARY OUTCOMES:
Cmax | 13 weeks
  Maximum blood drug concentration
Tmax | 13 weeks
  Peak time of blood drug concentration
BCVA | 13 weeks
  The best corrected visual acuity change
AUC0-t、AUCinf | 13 weeks
  The area under the plasma concentration time curves

CONTACTS AND LOCATIONS:
Overall Officials: xiu li zhao, doctor, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China